CLINICAL TRIAL: NCT03888547
Title: Integrating an Occupational Therapy Health and Wellness Program (OT-HAWP) Into an Existing Cancer Support Community
Brief Title: Integrating an Occupational Therapy Health and Wellness Program Into an Existing Cancer Support Community
Acronym: OT-HAWP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Indianapolis (Other)
Collaborators: Indiana Clinical and Translational Sciences Institute (Other)
Responsible Party: Principal Investigator, Katie M. Polo, DHS, OTR, CLT-LANA, Assistant Professor, University of Indianapolis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 0987
Record Dates: First submitted 2019-02-11; First posted 2019-03-25 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Cancer
Keywords: occupational therapy; health; wellness
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OT-HAWP (Experimental): The OT Health and Wellness Program will have four weeks of education and individual integration intervention modules:
  Week 1: Sleep Hygiene Week 2: Fatigue Management Week 3: Cancer-related cognitive impairments Week 4: Stress Management Each session will last 1.5 hours (45 minutes of group education and 45 minutes of individual modifications and strategy recommendations.
  Interventions: Other: Occupational Therapy Health & Wellness Education

INTERVENTIONS:
Other: Occupational Therapy Health & Wellness Education — The OT Health and Wellness Program will have four weeks of education and individual integration intervention modules. One of the investigators will lead each of these weekly modules under the direct supervision of the Principal Investigator. Investigators will be trained to provide the standardized educational module for each topic area and for using outcome measures. Each module will have an identified theme and information provided in each group will be education to topic, evidence based literature on intervention strategies, lifestyle, or environmental modifications that improve performance of daily activities that will last approximately 45 minutes. After, group sharing of ideas and individual identification of weekly goals for integration of 1-3 targeted interventions will occur and last approximately 30-45 minutes).

SUMMARY:
The number of cancer survivors today is growing exponentially and many survivors have unmet needs due to the late side effects of treatment. The purpose of this study is to explore the impact that a four-week Occupational Therapy Health and Wellness Program has on perceived satisfaction and performance of daily activities, fatigue, sleep quality, and health-related quality of life among adult community-dwelling cancer survivors.

Eligibility criteria for prospective participants includes cancer survivors with a past or present diagnosis that are at least 18 years old, able to consent, are English speaking, are able to fill out demographic information as well as pretest/posttest questionnaires, have indicated concerns within performance of daily activities and are able and willing to participate in a four-week Occupational Therapy Health and Wellness Program.

This quantitative study will use a prospective, one-group pretest-posttest design to explore the effects of a four-week Occupational Therapy Health and Wellness Program. Data that will be collected to track changes include physical, mental, and social health (measured by PROMIS questionnaire); fatigue levels (measured by the MAF questionnaire); Sleep quality (measured by the PSQI questionnaire); and self-perceived occupational performance and satisfaction (measured by the COPM interview/questionnaire) of community-dwelling cancer survivors.

Descriptive statistics will be used to compare pretest/posttest scores. Matched pairs t-test and Wilcoxin signed ranks test will be used if data is normally distributed. Normality will be tested by Shapiro wilks test and all data will be analyzed using t-tailed tests with significance set at .05.

DETAILED DESCRIPTION:
The purpose of this study is to explore the impact that a four-week Occupational Therapy (OT) Health and Wellness Program has on perceived satisfaction and performance of daily activities, fatigue, sleep quality, and health-related quality of life among adult community-dwelling cancer survivors.

The research questions for this study are as follows:

1. What changes occur in community-dwelling cancer survivors in Physical, Mental, and Social Health from the Patient-Reported Outcomes Measurement Information System (PROMIS) after a four-week Occupational Therapy Health and Wellness Program from initial pretest to posttest?
2. What changes occur in community-dwelling cancer survivors in self-perceived occupational performance and satisfaction from the Canadian Occupational Performance Measure (COPM) after a four-week Occupational Therapy Health and Wellness Program from initial pretest to posttest?
3. What changes occur in community-dwelling cancer survivors in fatigue from the Multidimensional Assessment of Fatigue Scale (MAF) after a four-week Occupational Therapy Health and Wellness Program from initial pretest to posttest?
4. What changes occur in community-dwelling cancer survivors in sleep quality from the Pittsburgh Sleep Quality Index (PSQI) after a four-week Occupational Therapy Health and Wellness Program from initial pretest to posttest? It is hypothesized that there will be improvements in participants self-perceived occupational performance and satisfaction, fatigue levels, sleep quality, as well their mental, physical, and social quality of life after participation in a four-week OT Health and Wellness Program. This study will explore occupational therapy health and wellness cancer programming in a new service setting of the community. It additionally will integrate innovative occupational therapy community cancer programming looking at called for participation outcomes.

METHODS This quasi-experimental study will use a single group pretest-posttest study design to explore the effects of a four-week Occupational Therapy Health and Wellness Program on physical, mental, and social health (PROMIS), fatigue levels (MAF), Sleep quality (PSQI), and self-perceived occupational performance and satisfaction (COPM) of community-dwelling cancer survivors.

Participants This study defines cancer survivor as any person who has been diagnosed with cancer from the time of diagnosis through the remainder of their life. Therefore, cancer survivors will be included irrespective of their phase of survivorship (i.e. actively receiving treatment, remission etc.).

An a priori power analysis using G*Power 3.1 was performed for a dependent-sample t test with the following parameters: two-tailed test, power of .80, a Type I error (α) of .05, and a medium effect size (d = .50). A minimum required sample size of 34 was determined. Taking into account attrition rate (25%), a target sample size is set for 43. Using results reported in a similar study of cancer survivors with an activity-based one week health program using the COPM, an effect size was calculated at .53 so the minimum sample size would be 30).

Data collected will be de-identified by using a participant code (first three letters of the participant's mother's first name and the last three digits of the participant's phone number). Participant IP addresses will not be collected in Qualtrics. A list of participant codes and their corresponding phone numbers will be stored on an encrypted google drive with access for investigators only in order to make reminder phone calls for meeting times. The study survey can be found at: https://uindy.co1.qualtrics.com/jfe/form/SV_56XfqHqrkLFYtNj

Procedures Recruitment. Survivors that are actively participating in programming at Cancer Support Communities Central Indiana location as well as their satellite facilities (Community Hospital, IU Health Simon Cancer Center, St. Vincent Cancer Care, and Hendricks Regional Health), and CSC community network partners (Little Red Door, Pink Ribbon etc.) will receive an informative flyer about the program. The program flyers will be posted at CSC and their satellite facilities as well as emailed to other community network partners for distribution. The OT Health and Wellness Program information will also be placed on CSC's programming schedule. Programming recruitment will also be through word from the investigators to their professional networks.

Screening. When a survivor calls to inquire about the OT programming, investigators will check if their results from the CSC Distress Screening Tool indicate the need for OT services. Those survivors that have indicated concerns of great severity on Cancer Support Community (CSC) Distress Screening Tool (Likert Items: very serious, serious, and moderately serious) in OT service provision areas related to finding meaning and purpose in life, disruptions in school/work/home life, fatigue, and sleep problems will be included in the study. This screening tool will be utilized to determine if participants are in need of the four-week OT Health and Wellness Program services and this data will be retained for the study.

Informed consent. Informed consent will happen at the survivor's first appointment with either the primary investigator or one of the co-investigators. Informed consent will be reviewed by one of the investigators and potential participants will indicate voluntary consent on Qualtrics. If the participants indicates voluntary consent to participate by continuing in Qualtrics, they will proceed into the COPM questionnaire. If the participant does not consent, it will take them out of Qualtrics. No data will be collected on those that do not provide voluntary consent.

Intervention. The OT Health and Wellness Program will have four weeks of education and individual integration intervention modules. One of the investigators will lead each of these weekly modules or students in the UIndy OTD program enrolled in OTD 620 Cancer Survivorship elective course will run the modules under the direct supervision of the Principal Investigator. Students will be trained to provide the standardized educational module for each topic area and will not be interacting with any study data. Each module will have an identified theme and information provided in each group will be education to topic, evidence based literature on intervention strategies, lifestyle, or environmental modifications that improve performance of daily activities that will last approximately 45 minutes. After, group sharing of ideas and individual identification of weekly goals for integration of 1-3 targeted interventions will occur and last approximately 30-45 minutes). The program will take place at CSC or one of their satellite facilities previously listed.

Data Analysis. Descriptive statistics will be used to describe the baseline and post-intervention characteristics of the sample. Nominal data will be presented as frequencies and percentages, while interval and ratio data will be reported as means and standard deviations or medians and interquartile ranges, dependent on whether the data are normally distributed. To determine if there is a significant difference in scores from pre-intervention to post-intervention, scores will compared using a paired t test, if the data are normally distributed, or the non-parametric Wilcoxon signed-ranks test if the data are not normally distributed. Normality will be determined using the Shapiro Wilk test. Data will be analyzed using IBM SPSS Statistics for Windows, Version 25.0. All comparisons will be two-tailed and a significance level of less than .05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Has present or past diagnosis of cancer
* Has indicated concerns affecting daily performance of activities, showing a need for OT programming
* Has access to Central Indiana Chapter of Cancer Support Community (CSC)
* Is able to consent
* Is able and willing to participate in demographic survey and pretest/posttest questionnaires
* Is able and willing to participate in a four-week Occupational Therapy Health and Wellness Program
* Is able to speak and understand English

Exclusion Criteria:

• Requires legal guardian to provide consent due to cognitive deficits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) change | pretest/post test: COPM will be collected at first intake appointment prior to the first OT-HAWP module and after the last OT-HAWP (4 weeks)
  Canadian Occupational Performance Measure (COPM) is a client centered outcome instrument that measures changes in a client's self-perception of occupational performance and satisfaction over time, and has been found to be a valid, reliable, and clinically useful outcome measure for occupational therapy research. In step two, the client is asked to rate the importance of each of the occupations to his/her life using a 10-point rating scale, the client is asked to use a 10 point scale to rate their own level of performance and satisfaction with performance for each of the five identified problems.
Patient-Reported Outcomes Measurement Information System-Global Health (PROMIS-G) | Change from baseline COPM to 4 weeks post
  Patient-Reported Outcomes Measurement Information System-Global Health (PROMIS-G) is an open access, person-centered questionnaire that measures physical, mental, and social health of adults, has been rigorously tested, has strong psychometric properties, and has cancer specific reference values. It is a 5 point likert scale.
Pittsburgh Sleep Quality Index (PSQI) change | Change from baseline PSQI to 4 weeks post
  Pittsburgh Sleep Quality Index (PSQI) is an open access, self-reported questionnaire that measures sleep quality and patterns in adults over a 1-month time interval, and has been found to be a reliable and valid assessment of sleep problems.
Multidimensional Assessment of Fatigue Scale (MAF) change | Change from baseline MAF to 4 weeks post
  Multidimensional Assessment of Fatigue Scale (MAF) is an open access, self-reported questionnaire that measures fatigue with recommended use in cancer rehabilitation.

CONTACTS AND LOCATIONS:
Overall Officials: Katie Polo, Principal Investigator — University of Indianapolis
Locations (1):
- Cancer Support Community, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Heinrich Heine (2013). *G Power 3 Software. Retrieved from: http://www.psycho.uni-duesseldorf.de/abteilungen/aap/gpower3/download-and-register.
- [Result] American Cancer Society (2018). Cancer Facts and Figures Retrieved from https://www.cancer.org/research/cancer-facts-statistics/all-cancer-facts-figures/cancer-facts-figures-2018.html
- [Result] Baxter MF, Newman R, Longpre SM, Polo KM. Occupational Therapy's Role in Cancer Survivorship as a Chronic Condition. Am J Occup Ther. 2017 May/Jun;71(3):7103090010P1-7103090010P7. doi: 10.5014/ajot.2017.713001. PMID 28422624
- [Result] Pergolotti M, Cutchin MP, Weinberger M, Meyer AM. Occupational therapy use by older adults with cancer. Am J Occup Ther. 2014 Sep-Oct;68(5):597-607. doi: 10.5014/ajot.2014.011791. PMID 25184473
- [Result] Polo KM, Smith C. Taking Our Seat at the Table: Community Cancer Survivorship. Am J Occup Ther. 2017 Mar/Apr;71(2):7102100010p1-7102100010p5. doi: 10.5014/ajot.2017.020693. PMID 28218583
- [Result] Hunter EG, Gibson RW, Arbesman M, D'Amico M. Systematic Review of Occupational Therapy and Adult Cancer Rehabilitation: Part 1. Impact of Physical Activity and Symptom Management Interventions. Am J Occup Ther. 2017 Mar/Apr;71(2):7102100030p1-7102100030p11. doi: 10.5014/ajot.2017.023564. PMID 28218585
- [Result] Carswell A, McColl MA, Baptiste S, Law M, Polatajko H, Pollock N. The Canadian Occupational Performance Measure: a research and clinical literature review. Can J Occup Ther. 2004 Oct;71(4):210-22. doi: 10.1177/000841740407100406. PMID 15586853
- [Result] Jensen RE, Potosky AL, Moinpour CM, Lobo T, Cella D, Hahn EA, Thissen D, Smith AW, Ahn J, Luta G, Reeve BB. United States Population-Based Estimates of Patient-Reported Outcomes Measurement Information System Symptom and Functional Status Reference Values for Individuals With Cancer. J Clin Oncol. 2017 Jun 10;35(17):1913-1920. doi: 10.1200/JCO.2016.71.4410. Epub 2017 Apr 20. PMID 28426375
- [Result] Grandner MA, Kripke DF, Yoon IY, Youngstedt SD. Criterion validity of the Pittsburgh Sleep Quality Index: Investigation in a non-clinical sample. Sleep Biol Rhythms. 2006 Jun;4(2):129-139. doi: 10.1111/j.1479-8425.2006.00207.x. Epub 2006 Jun 9. PMID 22822303
- [Result] Winstead-Fry P. Psychometric assessment of four fatigue scales with a sample of rural cancer patients. J Nurs Meas. 1998 Winter;6(2):111-22. PMID 10028778